CLINICAL TRIAL: NCT01724125
Title: An Electronic Personal Health Record for Mental Health Consumers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Benjamin Druss, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00012759; 1R18HS017829 (AHRQ)
Record Dates: First submitted 2012-04-25; First posted 2012-11-09 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Comorbid Conditions
Keywords: serious mental illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case (Experimental): Assigned a Personal Electronic Health Record
  Interventions: Other: personal electronic medical record
- Control: Usual Care (Active Comparator): Assigned to control arm, continued to receive care as usual in community. Was issued information on community health resources, but did not use research study personal health record.
  Interventions: Other: personal electronic medical record

INTERVENTIONS:
Other: personal electronic medical record

SUMMARY:
Electronic Personal Health Records (PHRs) hold promise in helping reshape healthcare by shifting the ownership and locus of health records from being scattered across multiple providers to an approach that is longitudinal and patient-centered. Given the complex health needs and the fragmentation of care for persons with serious mental illnesses, these individuals could derive particular benefit from a PHR. However, there are currently no established PHRs developed for use in this population.

In order to fill this gap, the investigators propose to develop, test, and disseminate a Personal Health Record for persons with serious mental illnesses and one or more comorbid medical condition. The Mental Health PHR (MH-PHR) builds on an established personal health record which was developed in partnership with medical consumers and is in wide use in a number of communities in the United States and abroad.

ELIGIBILITY:
Inclusion Criteria:

1. Currently in treatment at the CMHC.
2. Serious Mental Illness: based on or chart review;
3. One or more Chronic Medical Condition as ascertained via administrative records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Quality of Care | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Druss, MD MPH, Principal Investigator — Emory University
Locations (1):
- Grady Health Systems, Atlanta, Georgia, United States